CLINICAL TRIAL: NCT02375971
Title: RAINBOW Study: a Randomized, Controlled Study Evaluating the Efficacy and Safety of RAnibizumab Compared With Laser Therapy for the Treatment of INfants BOrn Prematurely With Retinopathy of Prematurity
Brief Title: RAINBOW Study: RAnibizumab Compared With Laser Therapy for the Treatment of INfants BOrn Prematurely With Retinopathy of Prematurity
Acronym: RAINBOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002H2301; 2014-003041-10 (EudraCT Number)
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Retinopathy of Prematurity
Keywords: intravitreal ranibizumab; laser ablation therapy; retinopathy of prematurity; preterm infants; RAINBOW
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ranibizumab 0.2 mg (Experimental): 1 intravitreal injection in both eyes on Day 1 (Baseline), with up to 2 re-treatments allowed for each eye if required
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.1 mg (Experimental): 1 intravitreal injection in both eyes on Day 1 (Baseline), with up to 2 re-treatments allowed for each eye if required
  Interventions: Drug: Ranibizumab
- Laser therapy (Active Comparator): Laser treatment to each eye on Day 1 (Baseline), with supplementary treatments allowed
  Interventions: Procedure: Laser therapy

INTERVENTIONS:
Drug: Ranibizumab — Administered as an intravitreal injection
  Arms: Ranibizumab 0.1 mg; Ranibizumab 0.2 mg
Procedure: Laser therapy — Transpupillary diode or frequency-doubled yttrium aluminum garnet (YAG) laser ablative therapy, following anesthesia or sedation
  Arms: Laser therapy

SUMMARY:
The purpose of this study was to determine if intravitreal ranibizumab is superior to laser ablation therapy in the treatment of retinopathy of prematurity (ROP).

DETAILED DESCRIPTION:
The study consisted of a screening period (screening and randomization could occur up to 3 days before the administration of the first investigational treatment), followed by a treatment and follow-up period (Day 1 to Day 169).

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with a birth weight of less than 1500 g
* bilateral ROP with one of the following retinal findings in each eye: Zone I, stage 1+, 2+, 3 or 3+ disease, or Zone II, stage 3+ disease, or Aggressive posterior retinopathy of prematurity (AP-ROP)

Exclusion Criteria:

* ROP disease characteristic in either eye other than that listed above at the time of the first investigational treatment
* A history of hypersensitivity (either the patient or the mother) to any of the investigational treatments or to drugs of similar chemical classes
* Had received any previous surgical or nonsurgical treatment for ROP (e.g., ablative laser therapy or cryotherapy, vitrectomy)
* Had been previously exposed to any intravitreal or systemic anti-VEGF agent (either the patient or the mother during this child's pregnancy)
* Had used (either the patient or the mother) other investigational drugs as part of another clinical study (other than vitamins and minerals) within 30 days or within 5 half-lives of the other investigational drug, whichever was longer
* Had ocular structural abnormalities that were assessed by the Investigator to have had a clinically significant impact on study assessments
* Had active ocular infection within 5 days before or on the day of first investigational treatment
* Had a history of hydrocephalus requiring treatment
* Had a history of any other neurological conditions that are assessed by the Investigator to have a significant risk of severe impact on visual function
* Had any other medical conditions or clinically significant comorbidities or personal circumstances that were assessed by the Investigator to have a clinically relevant impact on study participation, any of the study procedures, or on efficacy assessments (e.g., poor life expectancy, pupil not able to be adequately dilated, unable to comply with the visit schedule)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (83):
- United States (12):
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Morgantown, West Virginia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Ghent
- Croatia (2):
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Zagreb
- Czechia (3):
  - Novartis Investigative Site, Ostrava Poruba, Czech Republic
  - Novartis Investigative Site, Praha 4 - Podoli, Czech Republic
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Koebenhavn Ø, Denmark
- Novartis Investigative Site, Alexandria, Egypt
- Novartis Investigative Site, Tallinn, Estonia
- France (2):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Marseille
- Germany (2):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Hanover
- Greece (3):
  - Novartis Investigative Site, Ampelokipoi, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Goudi- Athens
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- India (6):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Vanchiyoor, Thiruvanantapuram
  - Novartis Investigative Site, New Delhi
- Italy (4):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Fiumicino, RM
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Yachiyo, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Zentsujichó, Kagawa-ken
  - Novartis Investigative Site, Shimajiri-Gun, Okinawa
  - Novartis Investigative Site, Izumi, Osaka
  - Novartis Investigative Site, Ohtsu-city, Shiga
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Sumida-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Novartis Investigative Site, Kaunas, LTU, Lithuania
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kota Kinabalu, Sabah
- Novartis Investigative Site, Querataro, Mexico
- Poland (2):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Wroclaw
- Romania (3):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Timișoara
- Russia (4):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Bratislava, Slovakia
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Eskişehir, Meselik
  - Novartis Investigative Site, Soguksu / Antalya, Turkey
  - Novartis Investigative Site, Zuhuratbaba / Istanbul, Turkey
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (3):
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Fleck BW, Reynolds JD, Zhu Q, Lepore D, Marlow N, Stahl A, Li J, Weisberger A, Fielder AR; RAINBOW Investigator Group. Time Course of Retinopathy of Prematurity Regression and Reactivation After Treatment with Ranibizumab or Laser in the RAINBOW Trial. Ophthalmol Retina. 2022 Jul;6(7):628-637. doi: 10.1016/j.oret.2022.02.006. Epub 2022 Feb 22. PMID 35202890
- [Derived] Stahl A, Lepore D, Fielder A, Fleck B, Reynolds JD, Chiang MF, Li J, Liew M, Maier R, Zhu Q, Marlow N. Ranibizumab versus laser therapy for the treatment of very low birthweight infants with retinopathy of prematurity (RAINBOW): an open-label randomised controlled trial. Lancet. 2019 Oct 26;394(10208):1551-1559. doi: 10.1016/S0140-6736(19)31344-3. Epub 2019 Sep 12. PMID 31522845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 87 sites: Austria(2), Belgium(2), Croatia(2), Czech Republic(3), Denmark(1), Egypt(1), Estonia(1), France(2), Germany(2), Greece(3), Hungary(2), India(6), Italy(4), Japan(17), Lithuania(1), Malaysia(2), Mexico(1), Poland(2), Romania(3), Russia(5), Saudi Arabia(1), Slovakia(1), Taiwan(2), Turkey(6), UK(3) and USA(12).
Pre-assignment Details: One patient was discontinued prior to receiving any study treatment and was later re-randomized; this patient is counted twice in the Randomized Set (FAS) (225). The number of unique participants randomized in the study is 224.
Period: Treatment (Day 1 - Baseline)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Started (All randomized patients to whom treatment had been assigned (FAS)) | 74 | 77 | 74
Safety Set (At least 1 application of investigational treatment and a 1 post baseline safety assessment) | 73 | 76 | 69
VEGF Set (All patients who provided valid Vascular endothelial growth factor (VEGF) plasma samples) | 19 | 26 | 51
PK Set (All patients who provided Pharmacokinetics (PK) serum samples) | 49 | 46 | 0
Completed (All patients who completed the treatment phase) | 73 | 76 | 69
Not Completed | 1 | 1 | 5
Not completed — Subj/Guardian Decision | 0 | 0 | 2
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Follow-Up Phase (up to Day 169)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Started (All patients who started the follow-up phase) | 73 | 76 | 69
Completed (All patients who completed the follow-up phase) | 66 | 71 | 64
Not Completed | 7 | 5 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Subject/Guardian Decision | 1 | 0 | 1
Not completed — Death | 4 | 4 | 4
Not completed — Withdrawal of Consent | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy | Total
Number analyzed (Participants) | 74 | 77 | 74 | 225
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational age at birth (weeks)
  Weeks | 25.8 (2.25) | 26.5 (2.57) | 26.2 (2.59) | 26.1 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 37 | 118
  Male | 33 | 37 | 37 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 27 | 22 | 23 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 3 | 7
  White | 43 | 45 | 45 | 133
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Absence of Active ROP and Absence of Unfavorable Structural Outcomes in Both Eyes at Week 24
Description: To achieve this outcome, patients must fulfill all the following criteria, 1) survival, 2) no intervention with a second modality for ROP, 3) absence of active ROP and 4) absence of unfavorable structural outcome. Retinopathy of prematurity (ROP) is a pathologic process that occurs in the incompletely vascularized, developing retina of low birth-weight preterm neonates.
Time Frame: Week 24
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 74 | 77 | 74
Percentage of Participants | 80.0 | 75.0 | 66.2
Statistical Analysis 1: Comparison: Ranibizumab 0.2 mg vs Ranibizumab 0.1 mg vs Laser Therapy; Test type: Superiority — The primary efficacy variable was treatment success, defined as the absence of active ROP and absence of unfavorable structural outcomes in both eyes 24 weeks after starting study treatment; p = 0.0254, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.9932 to 4.8235]

2. Secondary Outcome: Percentage of Participants Requiring Interventions With a Second Modality for ROP at Week 24
Description: Intervention for ROP in either eye at or before the 24-week assessment visit with a treatment modality other than the modality of the first study treatment. Only descriptive analysis done.
Time Frame: Week 24
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 74 | 77 | 74
Percentage of participants | 14.9 | 16.9 | 24.3

3. Secondary Outcome: Number of Participants Experiencing an Event, From the First Study Treatment to the Last Study Visit
Description: An event was defined as death, treatment switch, or the first occurrence of unfavorable structural outcomes in either eye. Only descriptive analysis done.
Time Frame: Day 1 (after initiation of study treatment) up to study exit (Day 169)
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 74 | 77 | 74
Participants | 14 | 18 | 23

4. Secondary Outcome: Percentage of Participants Having Recurrent ROP and Receiving Any Post-baseline Intervention at or Before Week 24
Description: Recurrence of ROP is defined as subjects receiving any post-baseline intervention in either eye at or before 24 weeks (ranibizumab re-treatment or switch to laser in the ranibizumab groups, switch to ranibizumab treatment in the laser group). Zone I consists of a circle, the radius of which extends from the center of the optic disc to twice the distance from the center of the optic disc to the center of the macula. Zone II extends centrifugally from the edge of zone I to the nasal ora serrata. Only descriptive analysis done.
Time Frame: Week 24
Population: The Full Analysis Set (FAS), which consisted of all participants with an observed value, was considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 74 | 77 | 74
Percentage of participants
  All participants | 31.1 | 31.2 | 18.9
  ZONE I | 35.7 | 53.3 | 28.6
  ZONE II | 28.3 | 17.4 | 13.0

5. Secondary Outcome: Percent of Participants With Ocular Adverse Events by Primary System Organ (SOCs) at Week 24
Description: Percent of Participants with Ocular Adverse Events regardless of Study Treatment and Procedure Relationship by Primary System Organ (SOCs) reported categorically (Mild, Moderate, Severe) 24 weeks after the first study treatment. Only descriptive analysis done.
Time Frame: Week 24
Population: The Safety Set was considered.
Measure: Number; unit: Percent of participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 73 | 76 | 69
Percent of participants
  Mild | 23.3 | 32.9 | 17.4
  Moderate | 4.1 | 6.6 | 13.0
  Severe | 2.7 | 1.3 | 2.9

6. Secondary Outcome: Mean Change in Ranibizumab Concentration in Pharmacokinetic Serum Samples Over Time at Day 1, Day 15 and Day 29
Description: Blood samples for the determination of ranibizumab concentrations were collected in the Ranibizumab treatment arms only at the following time points: within 24 hours after the first administration of ranibizumab, at Day 15 and at Day 29. Only descriptive analysis done.
Time Frame: Day 1 (Baseline), Day 15 and Day 29
Population: The PK Set, which consisted of all participants with at least one valid PK concentration value, was considered.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg
Number analyzed (Participants) | 49 | 46
picogram/milliliter (pg/mL)
  Day 1 (Baseline): number analyzed (Participants) | 43 | 43
  Day 1 (Baseline) | 24700.0 (52400.00) | 12100.0 (25500.0)
  Day 15: number analyzed (Participants) | 45 | 36
  Day 15 | 5830.0 (4750.0) | 27700.0 (144000)
  Day 29: number analyzed (Participants) | 31 | 24
  Day 29 | 1810.0 (2990.0) | 732.0 (535.0)

7. Secondary Outcome: Mean Change in Vascular Endothelial Growth Factor (VEGF) Levels Over Time at Day 1, Day 15 and Day 29
Description: Blood samples for the determination of systemic VEGF levels were collected at the following time points: before the first investigational treatment, at Day 15 and at Day 29. Only descriptive analysis done.
Time Frame: Day 1 (Baseline), Day 15 and Day 29
Population: The VEGF Set, which consisted of all participants with at least one valid VEGF concentration value, was considered.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 19 | 26 | 51
picogram/milliliter (pg/mL)
  Day 1: number analyzed (Participants) | 17 | 21 | 46
  Day 1 | 239.0 (226.0) | 230.0 (224.0) | 232.0 (240.0)
  Day 1 / no treatment modality switch: number analyzed (Participants) | 17 | 18 | 41
  Day 1 / no treatment modality switch | 239.0 (226.0) | 239.0 (233.0) | 233.0 (245.0)
  Day 15: number analyzed (Participants) | 15 | 26 | 44
  Day 15 | 466.0 (1500.0) | 118.0 (129.0) | 180.0 (214.0)
  Day 15 / no treatment modality switch: number analyzed (Participants) | 14 | 23 | 38
  Day 15 / no treatment modality switch | 498.0 (1560.0) | 124.0 (134.0) | 177.0 (224.0)
  Day 29: number analyzed (Participants) | 13 | 18 | 30
  Day 29 | 117.0 (84.0) | 176.0 (142.0) | 161.0 (132.0)
  Day 29 / no treatment modality switch: number analyzed (Participants) | 13 | 15 | 27
  Day 29 / no treatment modality switch | 117.0 (84.0) | 139.0 (75.3) | 163.0 (138.0)

8. Secondary Outcome: Total Number of Ranibizumab Injections Received at Week 24
Description: Patients randomized to receive Ranibizumab 0.1 mg or 0.2 mg received a single dose of intravitreal Ranibizumab to each eye on Day 1 (Baseline). Only descriptive analysis done.
Time Frame: Week 24
Population: The Safety Set was considered.
Measure: Number; unit: Injections
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 73 | 76 | 69
Injections | 73 | 76 | 13

9. Secondary Outcome: Percent of Participants With Non-Ocular Adverse Events by Primary System Organ (SOCs) at Week 24
Description: Percent of Participants with Non-Ocular Adverse Events regardless of Study Treatment and Procedure Relationship by Primary System Organ (SOCs) reported categorically (Mild, Moderate, Severe) 24 weeks after the first study treatment. Only descriptive analysis done.
Time Frame: Week 24
Population: The Safety Set was considered.
Measure: Number; unit: Percent of participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 73 | 76 | 69
Percent of participants
  Mild | 37.0 | 27.6 | 31.9
  Moderate | 24.7 | 34.2 | 27.5
  Severe | 23.3 | 19.7 | 17.4

10. Secondary Outcome: Mean Change From Baseline in Vital Signs (Body Length, Head Circumference and Knee to Heel Length) at Day 85 and Day 169
Description: Body Length, Head Circumference and Knee to Heel Length were assessed. Only descriptive analysis done.
Time Frame: Baseline, Day 85, Day 169
Population: The Safety Set was considered. Only patients with evaluable data at each time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 73 | 76 | 69
centimeter (cm)
  Day 85 / Body Length: number analyzed (Participants) | 61 | 63 | 60
  Day 85 / Body Length | 10.1 (2.59) | 11.0 (3.33) | 11.1 (3.65)
  Day 169 / Body Length: number analyzed (Participants) | 62 | 62 | 57
  Day 169 / Body Length | 18.7 (3.28) | 18.6 (3.66) | 19.0 (4.50)
  Day 85 / Head Circumference: number analyzed (Participants) | 62 | 62 | 59
  Day 85 / Head Circumference | 6.9 (1.96) | 6.5 (2.31) | 7.2 (2.13)
  Day 169 / Head Circumference: number analyzed (Participants) | 62 | 62 | 57
  Day 169 / Head Circumference | 10.4 (2.12) | 10.3 (2.56) | 10.6 (2.61)
  Day 85 / Knee to Heel Length: number analyzed (Participants) | 55 | 51 | 52
  Day 85 / Knee to Heel Length | 2.9 (1.90) | 3.1 (1.65) | 3.1 (2.02)
  Day 169 / Knee to Heel Length: number analyzed (Participants) | 53 | 52 | 52
  Day 169 / Knee to Heel Length | 5.4 (2.86) | 5.1 (2.19) | 5.3 (2.15)

11. Secondary Outcome: Mean Change From Baseline in Vital Signs (Weight) at Day 85 and Day 169
Description: Body weight was measured. Only descriptive analysis done.
Time Frame: Baseline, Day 85, Day 169
Population: The Safety Set was considered. Only patients with evaluable data at each time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 73 | 76 | 69
gram (g)
  Day 85 / Weight: number analyzed (Participants) | 63 | 66 | 60
  Day 85 / Weight | 2198.9 (615.68) | 2149.9 (754.27) | 2182.7 (612.70)
  Day 169 / Weight: number analyzed (Participants) | 62 | 62 | 60
  Day 169 / Weight | 3794.3 (782.48) | 3716.7 (897.15) | 3826.0 (882.17)

12. Secondary Outcome: Mean Change From Baseline in Vital Signs (Sitting Blood Pressure) at Day 85 and Day 169
Description: Blood Pressure measurements were not required by the protocol. Instead, the most recent Systolic and Diastolic Blood Pressure expressed in millimeters of mercury (mmHg) measured as part of the routine clinical care were used. Only descriptive analysis done.
Time Frame: Baseline, Day 85, Day 169
Population: The Safety Set was considered. Only patients with evaluable data at each time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 73 | 76 | 69
millimeters of mercury (mmHg)
  Day 85 / Sitting Diastolic Blood Pressure: number analyzed (Participants) | 47 | 46 | 41
  Day 85 / Sitting Diastolic Blood Pressure | 8.1 (14.66) | 7.0 (14.25) | 9.8 (16.95)
  Day 85 / Sitting Systolic Blood Pressure: number analyzed (Participants) | 47 | 46 | 41
  Day 85 / Sitting Systolic Blood Pressure | 6.3 (15.85) | 9.4 (15.73) | 15.5 (16.85)
  Day 169 / Sitting Diastolic Blood Pressure: number analyzed (Participants) | 45 | 46 | 40
  Day 169 / Sitting Diastolic Blood Pressure | 11.5 (15.60) | 11.8 (14.42) | 14.7 (17.05)
  Day 169 / Sitting Systolic Blood Pressure: number analyzed (Participants) | 45 | 46 | 40
  Day 169 / Sitting Systolic Blood Pressure | 10.2 (16.15) | 11.2 (13.45) | 17.7 (19.35)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit).
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- Laser: Laser treatment to each eye on Day 1 (Baseline), with supplementary treatments allowed
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser
All-Cause Mortality (participants affected / at risk) | 4/73 | 4/76 | 4/69
Serious Adverse Events (participants affected / at risk) | 26/73 | 24/76 | 24/69
Other Adverse Events (participants affected / at risk) | 43/73 | 47/76 | 37/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.2 mg (N=73) | Ranibizumab 0.1 mg (N=76) | Laser (N=69)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
Ileal atresia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 1 | 0
Retinopathy of prematurity (Eye disorders) | 2 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 2 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Cyst (General disorders) | 1 | 0 | 0
No adverse event (General disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 2 | 4 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Orbital infection (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Roseola (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 2
Septic shock (Infections and infestations) | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Greenstick fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Brain oedema (Nervous system disorders) | 2 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral cyst (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Perinatal brain damage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Breath holding (Psychiatric disorders) | 0 | 1 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dependence on oxygen therapy (Social circumstances) | 1 | 0 | 0
Haemodynamic instability (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.2 mg (N=73) | Ranibizumab 0.1 mg (N=76) | Laser (N=69)
Anaemia (Blood and lymphatic system disorders) | 4 | 8 | 5
Anaemia neonatal (Blood and lymphatic system disorders) | 2 | 4 | 1
Bradycardia (Cardiac disorders) | 2 | 5 | 1
Conjunctival haemorrhage (Eye disorders) | 6 | 6 | 2
Retinal haemorrhage (Eye disorders) | 6 | 10 | 7
Vitreous haemorrhage (Eye disorders) | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 5 | 4
Inguinal hernia (Gastrointestinal disorders) | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4 | 2
Pyrexia (General disorders) | 9 | 6 | 4
Conjunctivitis (Infections and infestations) | 1 | 6 | 2
Nasopharyngitis (Infections and infestations) | 7 | 5 | 4
Pneumonia (Infections and infestations) | 1 | 1 | 6
Rhinitis (Infections and infestations) | 3 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 2 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 8 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT02375971/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT02375971/SAP_003.pdf